CLINICAL TRIAL: NCT03869294
Title: Gemcitabine Plus S-1 as the First-line Chemotherapy in Chinese Patients With Advanced Pancreatic Cancer
Brief Title: GS Regimen as the First-line Chemotherapy in Chinese Advanced PC Patients
Status: Completed | Type: Observational
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Weijia Fang, MD, director, Zhejiang University
Other Study IDs: ZYYY-PAC1
Record Dates: First submitted 2019-03-08; First posted 2019-03-11 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Pancreatic Cancer; Chemotherapy Effect; Chemotherapeutic Toxicity
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- LAPC or MPC patients with GS first-line chemotherapy
  Interventions: Drug: GS

INTERVENTIONS:
Drug: GS — Gemcitabine plus S-1 (GS) was used to treat advanced pancreatic cancer

SUMMARY:
Gemcitabine plus S-1 (GS) prolonged progression-free survival (PFS) and greatly improved objective response rate (ORR) as well as disease control rate (DCR) of Asian patients with locally advanced and metastatic pancreatic cancer (PC). However, limited data of GS regimen exist on the efficacy and safety in the treatment of Chinese patients with advanced PC. To assess the efficacy and safety of gemcitabine plus S-1 (GS regimen) as the first-line chemotherapy in Chinese patients with advanced PC, we designed this prospective study.

ELIGIBILITY:
Inclusion Criteria:

* 1.Histologically confirmed pancreatic adenocarcinoma 2.Locally advanced or metastatic PC 3.Chemotherapy-naïve 4.ECOG performance status of 0 or 1 5. An adequate bone marrow, liver function and kidney function

Exclusion Criteria:

* 1.Age ≥80 years 2.Brain metastasis 3.With other malignancies 4.Chronic diarrhea, cardiac disease, pregnancy or breast feeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All advanced pancreatic cancer patients are diagnosed by histology to have pancreatic adenocarcinoma after a biopsy and received first-line GS chemotherapy at the Cancer Biotherapy Center of the First Affiliated Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | 2014-01-01 to 2017-12-31
  the time from the beginning of chemotherapy to the date of disease progression or death from any cause.
Overall survival | 2014-01-01 to 2017-12-31
  the time from the beginning of chemotherapy to the date of death from any cause.

SECONDARY OUTCOMES:
Objective response rate | 2014-01-01 to 2017-12-31
  the percentage of patients with CR or PR
adverse events | 2014-01-01 to 2017-12-31

CONTACTS AND LOCATIONS:
Locations (1):
- First affiliated hospital, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided